CLINICAL TRIAL: NCT00002620
Title: EFFECT OF DIBROMODULCITOL PLUS BCNU ON FREE INTERVAL AND SURVIVAL OF PATIENTS WITH SUPRATENTORIAL MALIGNANT BRAIN GLIOMAS, A PHASE III TYPE STUDY
Brief Title: Radiation Therapy in Treating Patients With Brain Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-26882; EORTC-26882
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Carmustine; Drug Therapy; Mitolactol

INTERVENTIONS:
Drug: carmustine
Drug: chemotherapy
Drug: mitolactol
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for patients with anaplastic astrocytomas.

PURPOSE: Randomized phase III trial to study the effectiveness of radiation therapy in treating patients with anaplastic astrocytomas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the disease-free interval and survival in patients with supratentorial malignant brain gliomas randomized to radiotherapy alone vs. radiotherapy plus radiosensitization with mitolactol (DBD) followed by DBD and carmustine.

OUTLINE: Randomized study. Group I: Radiotherapy. External-beam cranial irradiation with megavoltage equipment. Group II: Radiotherapy with Radiosensitization followed by Maintenance Chemotherapy. Radiotherapy as in Group I; with Mitolactol, DBD, NSC-104800; followed by DBD; Carmustine, BCNU, NSC-409962.

PROJECTED ACCRUAL: A total of 212 patients will be entered over more than 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed anaplastic astrocytoma Standard maximum resection or stereotactic biopsy required within 4 weeks prior to therapy

PATIENT CHARACTERISTICS: Age: Over 16 Performance status: ECOG/ZUBROD/WHO 0-2 Life expectancy: At least 8 weeks Hematopoietic: WBC greater than 4,000 Platelets greater than 100,000 Hematocrit greater than 30% Hepatic: Bilirubin less than 2 mg/dl Renal: Creatinine less than 1.5 mg/dl Creatinine clearance greater than 70 ml/min BUN less than 40 mg/dl Other: No major medical illness

PRIOR CONCURRENT THERAPY: No anticancer drugs between surgery and protocol treatment No steroids after 10 days following surgery (may be resumed occasionally during radiotherapy)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 1994-11; Primary Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Hildebrand, MD, Study Chair — Erasme University Hospital
Locations (14):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Belgium (4):
  - Hopital Universitaire Erasme, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels (Bruxelles)
  - Hopital Civil de Charleroi, Charleroi
  - Centre Hospitalier Regional de la Citadell, Liege (Luik)
- Neurologische Klinik der Henriettenstiftung, Hanover, Germany
- Regional Hospital Treviso, Treviso, Italy
- Netherlands (3):
  - Rotterdam Cancer Institute, Rotterdam
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Southampton General Hospital, Southampton, England

REFERENCES:
- [Result] Hildebrand J, Gorlia T, Kros JM, Afra D, Frenay M, Omuro A, Stupp R, Lacombe D, Allgeier A, van den Bent MJ; EORTC Brain Tumour Group investigators. Adjuvant dibromodulcitol and BCNU chemotherapy in anaplastic astrocytoma: results of a randomised European Organisation for Research and Treatment of Cancer phase III study (EORTC study 26882). Eur J Cancer. 2008 Jun;44(9):1210-6. doi: 10.1016/j.ejca.2007.12.005. Epub 2008 Jan 14. PMID 18248979
- [Result] Hildebrand J, Sahmoud T, Mignolet F, Brucher JM, Afra D. Adjuvant therapy with dibromodulcitol and BCNU increases survival of adults with malignant gliomas. EORTC Brain Tumor Group. Neurology. 1994 Aug;44(8):1479-83. doi: 10.1212/wnl.44.8.1479. PMID 8058153